CLINICAL TRIAL: NCT06546007
Title: Clinical Study To Evaluate the Sensitivity of Circulating Iset® by Rarecells Molecular Biomarkers for Early Detection of Lung Cancer
Brief Title: Rarecells Molecular Biomarkers for Early Detection of Lung Cancer
Acronym: BioMolCTC
Status: Recruiting | Type: Observational
Sponsor: Rarecells Diagnostics SAS (Industry)
Collaborators: Meditrial Europe Ltd. (Industry); Meditrial SrL (Industry)
Responsible Party: Sponsor
Other Study IDs: BIOMOLCTC-24-01
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer; Pulmonary Neoplasm
Keywords: Circulating tumor cells; Lung cancer; Circulating tumor DNA; Pulmonary neoplasm
MeSH Terms: conditions — Lung Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Analysis of tumor DNA (CTC-DNA) in blood samples from subjects with lung cancer undergoing lung surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patient with early lung cancer: Patients with a diagnosis of lung cancer, planned for lung resection with curative intent.
  Interventions: Diagnostic Test: CTC-DNA

INTERVENTIONS:
Diagnostic Test: CTC-DNA — ctDNA for the analysis of lung cancer mutations in patients with operable tumors.
  Other Names: ctDNA

SUMMARY:
Early diagnosis of lung cancer is a public health priority. Additionally, early detection of recurrences after treatment is crucial for optimizing disease management.

This study seeks to demonstrate the accuracy of the Rarecells ISET® circulating tumor cells DNA (CTC-DNA), combined with circulating tumor DNA (ctDNA), for the early diagnosis of lung cancer.

DETAILED DESCRIPTION:
Researching for tumor biomarkers in the blood, circulating tumor cells (CTCs), and circulating tumor DNA (ctDNA) can non-invasively detect signs of cancer without risk to the patient. These are ideal and risk-free methods for monitoring patients and early detection of lung cancer.

This study aims to assess the sensitivity of molecular analyses performed on circulating tumor DNA in the blood and on DNA from circulating tumor cells, isolated using the highly sensitive ISET® method. The purpose is to assess two circulating molecular biomarkers in the field of liquid biopsy in patients with lung cancer: Rarecells ISET® CTC-DNA and ctDNA.

Subjects eligible for inclusion in the study are individuals diagnosed with operable lung cancer who will undergo biopsy or surgical resection of the tumor. Upon enrolment in the trial, participants will undergo an assessment including low-dose CT scan, isolation of CTCs by the ISET® method, and separation of plasma for analysis of ctDNA.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged between 35 and 85 years
2. Patient diagnosed with resectable lung cancer (by imaging and/or pathological examination) not yet treated for this cancer.
3. Patient capable of giving free, informed, and express consent

The assessment of successful elected surgery implies, but is not limited to, the following:

* Exclusion of detectable extra thoracic and distant metastases
* Determination of the presence or absence of superior mediastinal lymph node metastases
* Definition of the histologic or cell type, whenever possible
* Evaluation of operative risk

Exclusion Criteria:

1. Patient diagnosed and/or treated previously for lung cancer or another cancer, regardless of duration
2. Patient treated with neoadjuvant treatment
3. Pregnant women
4. Patient presenting psychiatric or neurological disorders preventing them from understanding the research

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of lung cancer, planned for lung resection with curative intent.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Comparative and complementary in operable patients diagnosed with cancer | 30 days post procedure
  Number of patients with lung cancer-related mutations by CTCDNA alone, by ctDNA alone and by the ctDNA -CTCDNA pair divided by the number of patients with cancer enrolled in the study

SECONDARY OUTCOMES:
Comparative and complementary sensitivity of CTC-DNA and ctDNA per histological subtype | 30 days post procedure
  Number of patients with lung cancer-related mutations by CTCDNA alone, by ctDNA alone and by the ctDNA -CTCDNA pair per histologic subtype

CONTACTS AND LOCATIONS:
Overall Officials: Patrizia Paterlini, MD, PhD, Study Director — Rarecells
Locations (1):
- Università Cattolica del Sacro Cuore Gemelli Hospital, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Rarecells - sponsor website — http://www.rarecells.com
- See also: Meditrial Contract Research Organization Website — http://www.meditrial.net